CLINICAL TRIAL: NCT04093349
Title: Phase 1/2, Dose-escalation Study to Evaluate the Safety, Tolerability and Efficacy of a Single Intravenous Infusion of SPK-3006 in Adults With Late-onset Pompe Disease
Brief Title: A Gene Transfer Study for Late-Onset Pompe Disease (RESOLUTE)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPK-3006-101; 2019-001283-30 (EudraCT Number)
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Pompe Disease; Pompe Disease (Late-onset); Glycogen Storage Disease Type 2; Glycogen Storage Disease Type II; LOPD; Lysosomal Storage Diseases; Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPK-3006 (Experimental): All participants who meet the eligibility criteria will receive a single intravenous (i.v.) administration of SPK-3006.
  Interventions: Genetic: SPK-3006

INTERVENTIONS:
Genetic: SPK-3006 — adeno-associated viral (AAV) vector

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of a single intravenous infusion of SPK-3006 in adults with clinically moderate, late-onset Pompe disease receiving enzyme replacement therapy (ERT). Participants will be treated in sequential, dose-level cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Males and Females ≥18 years of age with late-onset Pompe disease;
* Received ERT for at least the previous 24 months
* Have clinically moderate, late-onset Pompe disease characteristics;
* Agree to use reliable contraception.

Exclusion Criteria:

* Active hepatitis B and/or C;
* Significant underlying liver disease;
* Human immunodeficiency virus (HIV) infection;
* Prior hypersensitivity to rhGAA;
* Pre-existing anti-AAV neutralizing antibody titers;
* High titer antibody responses to rhGAA;
* Requires any invasive ventilation or requires noninvasive ventilation while awake and upright;
* Received any prior vector or gene transfer agent;
* Active malignancy (except non-melanoma skin cancer);
* History of liver cancer;
* Pregnant or nursing women;
* Any evidence of active infection at the time of SPK-3006 infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2032-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Number of adverse and serious adverse events (AEs/SAEs), including clinically significant abnormal laboratory values. | Up to 5 years
  Adverse events.
Occurrence of immune response against AAV capsid | Up to 5 years
Occurrence of immune response against GAA transgene | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tahseen Mozaffar, MD, Principal Investigator — University of California Irvine Health
Locations (29):
- United States (10):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California Irvine Health, Orange, California
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research & Treatment Center, Fairfax, Virginia
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - Montreal Neurological Hospital, Montreal, Quebec
- Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - CHU Paris IdF Ouest - Hôpital Raymond Poincaré, Garches
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Assistance Publique Hôpitaux de Marseille, Marseille
  - Nice University Hospital, Nice
- Friedrich-Baur-Institut Neurologische Klinik Ludwig-Maximilians-Universität München, München, Germany
- Italy (5):
  - Universita Degli Studi Di Messina - Dipartimento di Medicina Clinica e Sperimentale, Messina
  - Universita Degli Studi Di Milano, Laboratorio di Biochimica e Genetica della Malattie Neuromuscolari, Milan
  - Malattie Metaboliche Universita Degli Studi Di Napoli Federico II, Naples
  - UO Neurologia Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda Ospedaliera Universitaria Città della Salute e della Scienza di Torino - Neurology, Osp. Molinette, Torino
- Erasmus Medical Center, Rotterdam, Netherlands
- United Kingdom (3):
  - New Queen Elizabeth Hospital Birmingham, Birmingham, GBR
  - The Royal Free London NHS Foundation Trust, London, GBR
  - Salford Royal MHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No